CLINICAL TRIAL: NCT00209807
Title: Effect of Escitalopram vs. Reboxetine on Somatic and Visceral Sensitivity of Patients With Major Depressive Disorder: a Randomized, Double Blind Clinical Trial
Brief Title: Effect of Escitalopram vs. Reboxetine on Gastro-intestinal Sensitivity of Patients With Major Depressive Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Miguel Casas Brugué, Servei de Psiquiatria. Hospital Universitari Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PFD-ESC
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Major Depression; Pain; Abdominal Pain
Keywords: major depression; pain; escitalopram; reboxetine; visceral sensitivity; somatic sensitivity
MeSH Terms: conditions — Depressive Disorder, Major; Pain; Abdominal Pain | interventions — Escitalopram; Reboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): subjects with MDD randomized to Escitalopram
  Interventions: Drug: escitalopram
- 2 (Active Comparator): MDD patients receiving reboxetine
  Interventions: Drug: Reboxetine
- 3 (Other): Healthy volonteers
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: escitalopram — escitalopram 10 mg/d for 6 weeks
  Other Names: reboxetine
  Arms: 1
Drug: Reboxetine — Reboxetine 8 mg/d for 6 weeks
  Arms: 2
Other: No intervention — This group of healthy volonteers will receive no drug and will be a healthy comparator.
  Arms: 3

SUMMARY:
Patients with major depressive disorder (MDD) commonly have many gastrointestinal complaints. Gastrointestinal pain is classified into 2 categories: visceral and somatic pain. The main aim of this study is to compare somatic and visceral sensitivity between healthy people and pateints with MDD. These two sensitivities will be assessed by the 2 following tests: standardized rectal distension and Transdermal transcutaneous electric nerve stimulation. Thereafter, patients with MDD will be randomly allocated to escitalopram or reboxetine. After 6 weeks of treatment, somatic and visceral sensitivity will be reassessed.

ELIGIBILITY:
Inclusion Criteria:

* MDD according with DSM-IV-TR
* Hamilton depression scale > 21

Exclusion Criteria:

* history of gastrointestinal illness
* history of escitalopram, citalopram or reboxetine allergy.
* history of escitalopram, citalopram or reboxetine resistant depression.
* other axis I psychiatric disorder.
* a punctuation > 2 on the suicide item of the Ham-D.
* history of ECT during the past 6 months.
* pharmacological failure of the present depressive episode.
* pregnancy or nursing.
* treatment with drugs that may interact with study medication.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2005-09; Primary Completion 2009-06 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
rectal distension Transcutaneous Electrical Neuro-Stimulation | 1-7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Casas Miguel, Prof., Principal Investigator — Hospital Universitari Vall d'Hebron Research Institute
Locations (1):
- Hospital Universitari vall d'Hebron, Barcelona, Catalonia, Spain